CLINICAL TRIAL: NCT04032548
Title: Comparison of Effectiveness of Propolis Mouthwash on Gingivitis - Randomized Controlled Clinical Study
Brief Title: Effectiveness of Propolis Mouthwash on Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Shilpa Gunjal, Associate Professor, Mahsa University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RP104-10/16
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects were asked to rinse 10 ml of mouthwash twice daily for 21 days.
  Interventions: Drug: Placebo mouthwash
- Propolis (Experimental): Subjects were asked to rinse 10 ml of mouthwash twice daily for 21 days.
  Interventions: Drug: Propolis mouthwash
- Chlorhexidine (Active Comparator): Subjects were asked to rinse 10 ml of mouthwash twice daily for 21 days.
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Placebo mouthwash — After using mouthwash for 21 days, they are instructed to refrain from mouthwash for 14 days (wash out period).
  Other Names: Mouthwash
  Arms: Placebo
Drug: Propolis mouthwash — After using mouthwash for 21 days, they are instructed to refrain from mouthwash for 14 days (wash out period).
  Other Names: Mouthwash
  Arms: Propolis
Drug: Chlorhexidine mouthwash — After using mouthwash for 21 days, they are instructed to refrain from mouthwash for 14 days (wash out period).
  Other Names: Mouthwash
  Arms: Chlorhexidine

SUMMARY:
Mouthrinses have been in used for centuries as breath fresheners, medicaments, and antiseptics. Recently, propolis has caught the eyes of dentists worldwide and researches are being carried out to infuse the usage of propolis in the dental health care treatments. There is belief that propolis may have a role as a tooth decay prophylaxis and help heal oral ulcers. Propolis is used as mouthwash, toothpaste, oral gel, and throat lozenges because of its proclaimed antibacterial and anti-inflammatory properties. Propolis has shown activity against common periodontal microorganisms, such as Candida species and the Streptococci mutans in vitro studies. Till date, no study has evaluated the clinical and microbiological effects of Malaysian Propolis as a mouthwash. Thus, the present study is designed to evaluate the effectiveness of Propolis as a mouthwash in the reduction of Plaque and gingivitis.The aim of the study is to assess and compare the effectiveness of Propolis mouthrinse with Chlorhexidine mouthrinse.

DETAILED DESCRIPTION:
The Randomized Controlled Clinical study with latin-square cross-over design would be used to assess and compare the effectiveness of Propolis and Chlorhexidine mouthrinse on gingivitis. Subjects with chronic generalized gingivitis with age group of 18-30 years will be selected for the study as the target population. Subjects who meet the inclusion and exclusion criteria will be selected and screened for the plaque and gingival status before including them in the study. They will be randomly divided into three groups.

Group 1: 15 subjects (Placebo mouthwash) Group 2: 15 subjects (Propolis mouthwash) Group 3: 15 subjects (Chlorhexidine mouthwash)

ELIGIBILITY:
Inclusion Criteria:

* Gingival index >1
* Periodontal pocket depth ≤ 3 mm
* Clinical attachment loss "0"
* Provision of written informed consent
* Good systemic health.

Exclusion Criteria:

* Severe periodontal disease, as characterized by purulent exudates, generalized mobility, and/or severe recession
* Any condition that requires antibiotic premedication for the administration of a dental prophylaxis.
* Self-reported pregnancy, intent to become pregnant during the study, or breast-feeding.
* Any diseases or condition that could be expected to interfere with the safe completion of the study.
* History of antibiotic use in the previous 3 months.
* Individuals with orthodontic appliances or prosthetic appliances that would interfere with evaluation.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Gingival Index (GI) | Difference for the mean gingival score from baseline to 21 days.
  The primary outcome variable was the differences for the mean gingival score from baseline to 21 days.
  The gingival index ranges from 0-3 which is a continuous scale. '0' indicates normal healthy gingiva without inflammation (better score) ; and score '3' indicates severe gingival inflammation (worst score).
  The index teeth of each participant were examined and gingival status is scored. The score for each subject is added and divided by the total number of teeth examined.
  The average/mean gingival score obtained from each subject is added for all the subjects and divided by the total number of participants. Higher score indicates worst score.
Change in Plaque Index (PI) | Difference in the mean reduction of Plaque score from baseline to 21 days.
  The primary outcome variable was the differences for the mean plaque score from baseline to 21 days.
  The plaque index ranges from 0-3 which is a continuous scale. '0' indicates no plaque on teeth (better score) ; and score '3' indicates abundance of plaque on the teeth (worst score).
  The index teeth of each participant were examined and plaque score is recorded. The score for each subject is added and divided by the total number of teeth examined.
  The average/mean plaque score obtained from each subject is added for all the subjects and divided by the total number of participants. Higher score indicates worst score.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Gunjal, Ph.D, Principal Investigator — Mahsa University
Locations (1):
- Shilpa, Jenjarum, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunjal S, Pateel DGS. Comparative effectiveness of Propolis with chlorhexidine mouthwash on gingivitis - a randomized controlled clinical study. BMC Complement Med Ther. 2024 Apr 6;24(1):154. doi: 10.1186/s12906-024-04456-8. PMID 38582863